CLINICAL TRIAL: NCT01877694
Title: A Multicenter, Randomized Study of the Efficacy and Safety of Auriclosene (NVC-422) Ophthalmic Solution 0.3% for the Treatment of Bacterial Conjunctivitis
Brief Title: Efficacy and Safety of Auriclosene (NVC-422) in the Treatment of Bacterial Conjunctivitis
Acronym: BACTOvation™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaBay Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL1301
Record Dates: First submitted 2013-06-07; First posted 2013-06-14 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Bacterial Conjunctivitis
Keywords: pink eye
MeSH Terms: conditions — Conjunctivitis, Bacterial; Conjunctivitis | interventions — NVC-422

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auriclosene Solution 0.3% (Experimental): Dosed QID for 4 Days
  Interventions: Drug: Auriclosene Solution 0.3%
- Auriclosene Vehicle (Placebo Comparator): Dosed QID for 4 days
  Interventions: Drug: Auriclosene Vehicle

INTERVENTIONS:
Drug: Auriclosene Solution 0.3% — Ophthalmic solution dispensed as drops onto the eye
  Other Names: NVC-422
  Arms: Auriclosene Solution 0.3%
Drug: Auriclosene Vehicle — Ophthalmic Vehicle solution dispensed as drops onto the eye
  Arms: Auriclosene Vehicle

SUMMARY:
The purpose of this study is to evaluate the microbiological and clinical efficacy of Auriclosene compared to its vehicle for bacterial conjunctivitis. Adults and children one year of age and older with bacterial conjunctivitis in at least one eye may be eligible. Subjects will be randomly assigned to receive either Auriclosene Ophthalmic Solution or Vehicle Ophthalmic Solution.

DETAILED DESCRIPTION:
This is a randomized (1:1) double-masked, vehicle-controlled, multi-center, parallel group study with two treatment arms: Auriclosene Ophthalmic Solution 0.3% ("Auriclosene") and Auriclosene Vehicle ("Vehicle").

Subjects that meet all inclusion/exclusion criteria will be enrolled into the study, randomized and evaluated at 3 visits:

* Visit 1: Screening, Day 1
* Visit 2: Day 3 (±1)
* Visit 3: Day 5 (+1) Test of Cure/Exit

IP will be dosed OU (both eyes) QID for 4 days. Microbiological specimens will be collected from each eye at each visit.

Visual Acuity will be assessed OU at each visit as well as rating of the ocular signs: lid erythema and swelling, bulbar and palpebralconjunctival injection, and conjunctival discharge/exudate.

ELIGIBILITY:
Inclusion Criteria:

* 1 year of age and older
* Bulbar conjunctival injection
* Conjunctival discharge/exudate
* Signs and symptoms of bacterial conjunctivitis in at least one eye for 3 days or less
* Other inclusion criteria per protocol

Exclusion Criteria:

* Suspected fungal, viral, Chlamydia or Acanthamoeba co-infection based on clinical diagnosis
* Any drug treatment in either eye for the current episode of bacterial conjunctivitis prior to study enrollment
* Other exclusion criteria per protocol

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Microbiological Success | 5 days
  Eradication of all pre-therapy isolates

SECONDARY OUTCOMES:
Clinical Cure | 5 days
  Resolution of all signs and symptoms

OTHER OUTCOMES:
Resolution of individual ocular signs and symptoms | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: David W. Stroman, Ph.D., Study Director — NovaBay Pharmaceuticals, Inc.
Locations (21):
- United States (21):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Anaheim, California
  - Bellflower, California
  - Glendale, California
  - Huntington Beach, California
  - Clearwater, Florida
  - Woodstock, Georgia
  - Evansville, Indiana
  - Newton, Kansas
  - Whitehouse Station, New Jersey
  - Huntersville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Corsicana, Texas
  - San Antonio, Texas
  - Clinton, Utah
  - Charlottesville, Virginia
  - Midlothian, Virginia
  - Spokane, Washington

REFERENCES:
- [Derived] Lee CS, Lee AY, Akileswaran L, Stroman D, Najafi-Tagol K, Kleiboeker S, Chodosh J, Magaret A, Wald A, Van Gelder RN; BAYnovation Study Group. Determinants of Outcomes of Adenoviral Keratoconjunctivitis. Ophthalmology. 2018 Sep;125(9):1344-1353. doi: 10.1016/j.ophtha.2018.02.016. Epub 2018 Mar 27. PMID 29602567